CLINICAL TRIAL: NCT03089788
Title: Methodological Study to Compare the Effect of Different Methods of Measuring Cat Allergy Symptoms in Patients That Have Immunized Their Cats With FEL-CMV.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Thomas Kuendig, Prof. Dr. med, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZU-HypoCat-002
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based test and skin test (Other)
  Interventions: Other: Home-based test; Other: Skin test

INTERVENTIONS:
Other: Home-based test — Home-based tests in which the participant pets his/her cat until he/she reaches a certain symptom strength.
Other: Skin test — Skin Prick Tests will be performed with registered cat allergen extract.

SUMMARY:
In this Project we will monitor the symptoms of cat allergic participants who live together with a cat which is immunized with FEL-CMV using the novel symptom recording method "HypoScore", a General weekly symptom score, and a skin prick test before and after immunization of the cat. This project may enable us to determine if the scoring System and the tests are able to detect a difference in participant symptoms before and after immunization of the cats.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent after participants' information
* 18 to 65 years, male or female
* Participant understands the nature, meaning and scope of the study
* Positive screening prick test (wheal diameter ≥ 3mm) to Histamine dihydrochloride 10mg/ml
* Positive screening prick test (mean wheal diameter ≥ 3 mm) when tested with already standardized cat allergen extract
* Positive screening scratch test when tested with cat dander sample of participant's cat.
* Living with a cat in the same household and parallel participation in the cat study in which the cat will be immunized
* A positive clinical history with inhalant allergy presumably due to cat allergen

Exclusion Criteria:

* Immunosuppression or haematological diseases, in particular anaemias or leukaemia
* Other previous or current condition or participation in clinical trials influencing the results of the present study by discretion of the investigator
* Incapable of understanding the nature, meaning or scope of the research project or incapable of giving written informed consent
* Unwilling or incapable of following the study procedures, e.g. due to language problems, psychological disorders, dementia, known or suspected drug or alcohol abuse etc.
* Women who are pregnant or breast feeding or having the intention to become pregnant during the course of the study
* Positive skin reaction in the screening prick test to negative control
* History of anaphylactic reaction to pet allergens
* Severe diseases influencing the results of the present study by discretion of the investigator
* Immunotherapy with Fel d 1 / cat allergen preparation during the past two years.
* Skin lesions and excessive hair growth in the skin test areas
* Treatment with prohibited concomitant medications with the exception of medications with local effects which will not influence the results of the skin tests and the results of the other tests (testing period)
* The participant should not suffer from other respiratory allergies during this study (people who suffer from asthma are not excluded)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Organ specific symptom sum score of HypoScore measured after petting the cat at baseline versus week 24 | Comparison of the symptom score of 3 baseline measurements and measurement in week 24
  Organ specific symtpom score component of HypoScore is measured with a questionnaire before and after the participants perform the tests with their cats (petting the cat until certain symptoms are reached).
General weekly symptom score measured at baseline (with unimmunized cat) versus week 24 (with immunized cat) | Measured over 25 weeks
  General weekly symptom score is measured with a weekly questionnaire. This questionnaire will be filled in on a weekly Basis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No